CLINICAL TRIAL: NCT03144401
Title: Preoperative vs. Postoperative Misoprostol in Elective Cesarean Section: A Double-blind Randomized Clinical Trial
Brief Title: Preoperative vs. Postoperative Misoprostol in Elective Cesarean Section
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed S Sweed, MD, Assistant Professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AS1374
Record Dates: First submitted 2017-04-29; First posted 2017-05-08 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Cesarean Section
Keywords: cesarean section; Misoprostol; sublingual; uterotonics
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Preoperative (Active Comparator): • Group no.1 will receive preoperative sublingual 400 microgram of misoprostol (Sigma) "2 tablets" and postoperative sublingual placebo"2 tablets".
  Interventions: Drug: Misoprostol; Other: Placebo
- Postoperative (Active Comparator): • Group no.2 will receive preoperative sublingual placebo "2 tablets" and postoperative sublingual 400 microgram of misoprostol (Sigma) " 2 tablets" .
  Interventions: Drug: Misoprostol; Other: Placebo

INTERVENTIONS:
Drug: Misoprostol — mesotac
Other: Placebo — Placebo tablet identical to the misoprostol tablet but without the active ingredient

SUMMARY:
This prospective double-blind placebo-controlled randomized clinical trial will be conducted at Ain-Shams University Maternity Hospital from April 2017 till October 2017. 120 women candidate foe elective cesarean section will receive preoperative sublingual 400 microgram of misoprostol, and another 120 women will receive postoperative sublingual 400 microgram of misoprostol.

ELIGIBILITY:
Inclusion Criteria:

* Patients booked for elective cesarean section.
* Singleton pregnancies.
* Full term pregnancies (GA 37- 42 Wks).
* Age (18-40 yrs).
* body mass index (BMI) (20-30(Kg/m2 .

Exclusion Criteria:

* Contraindication to spinal anesthesia.
* Blood dyscrasias.
* Large fibroids.
* Multiple pregnancies.
* Overdistended uterus eg. Hydramnios.
* Pre-eclampsia.
* Marked maternal anemia (Preoperative hemoglobin < 9 gm/dl).
* Previous history of PPH.
* Contraindications to prostaglandin therapy (e.g. history of severe bronchial asthma or allergy to misoprostol.
* Placenta previa.
* Previous myomectomy.
* Extreme of BMI (<20 or >30 Kg/m2 ).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2018-01-12 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Need for extra uterotonics | 24 hours

SECONDARY OUTCOMES:
intraoperative blood loss | intraoperative
postpartum hemorrhage | 24 hours
neonatal outcome | 5 minutes
  measured by APGAR score at 1 and 5 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt